CLINICAL TRIAL: NCT06683196
Title: The Effects of Scapular Taping Techniques on Grip Strength and Hand Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Eda AKBAŞ, Associate Professor, Zonguldak Bulent Ecevit University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BEUN-2024/18-09
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-10

CONDITIONS: Grip Strength; Hand Function
Keywords: grip strength; hand function; taping; scapular taping

STUDY DESIGN:
Intervention Model Description: On three different days, each participant will receive taping with one of the three tape types (Kinesiotape, Rigid Tape and Placebo Tape ). This approach aims to prevent fatigue and habituation during evaluations. To minimize potential bias in measurements, the sequence of tape types will be changed across the three days.
Masking Description: The researcher who will evaluate the patients after taping will not know which group the patients are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Group (Experimental): All interventions applied to all of the participants.
  Interventions: Other: Kinesio Taping; Other: Rigid Taping

INTERVENTIONS:
Other: Kinesio Taping — 3 types of taping (kinesiotape, rigid tape and placebo tape) applied to all participants.
Other: Rigid Taping — 3 types of taping (kinesiotape, rigid tape and placebo tape) applied to all participants.

SUMMARY:
This study aims to investigate the effects of different types of taping applied to the scapular region on grip strength and hand function.

DETAILED DESCRIPTION:
Disorders in the alignment of the scapula can lead to mechanical disorders in the proximal. This can lead to a decrease in proximal stability and a negative effect on force production in the distal.

Kinesio tape can stimulate mechanoreceptors through the skin with applied tension, create positional awareness, improve fascia alignment and reduce edema. It is also used to lift soft tissues in areas with pain and inflammation or to limit and increase movement. Rigid taping is performed using non-elastic material and is preferred to increase stabilization and prevent injuries . There are also studies showing that rigid tape increases sensorimotor and proprioceptive senses ).

In a study it was shown that kinesio taping applied to the scapular region improved upper extremity function. In a studyi, it was found that taping improved function in those with lumbar radiculopathy and that elastic taping was more effective than rigid taping. Although there are studies comparing kinesio taping and rigid taping on shoulder joint range of motion and muscle strength, there is no study examining the effects of different tapings applied to the scapular region on grip strength and hand function. In addition, the positive effects of shoulder stabilization exercises on hand skills and grip strength have been shown in the literature.

Studies examining taping and hand functions have generally focused on the forearm and finger areas. The relationship between interventions in the scapular region and grip strength and function has not been sufficiently investigated in the literature, and filling this gap is important for functional rehabilitation.

Previous studies have indicated that taping is effective in injuries affecting the scapular region and upper extremity. This study will examine the effects of different types of taping applied to the scapular region on grip strength and hand function.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 25,
* With undamaged skin tissue in the area where taping will be applied,
* Who are willing to participate in the study.

Exclusion Criteria:

* Individuals with a pathology, disease, or disability affecting upper extremity function,
* Who have experienced trauma/surgery affecting motor and sensory function in the upper extremity and neck region within the last 6 months,
* Who have normal joint motion limitations in the neck, shoulder, elbow, hand, and wrist joints,
* Who have received corticosteroid treatment in the shoulder region within the last 3 months,
* Who have received physiotherapy within the last 3 months.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Pinch Grip Strength | 7 days
  For pinch grip strength measurement, a mechanical pinch meter (Baseline®, USA) will be used. Lateral (key) pinch, two-point (bipod, tip) pinch, and three-point (tripod, palmar) pinch measurements will be performed separately. For the lateral pinch, the patient will be asked to squeeze the end of the pinch meter between the thumb and the lateral surface of the middle phalanx of the second finger with maximum force. For the two-point pinch strength measurement, the patient will be asked to squeeze the pinch meter between the thumb and the pulp of the second finger, and for the three-point pinch strength measurement, between the thumb, the second finger, and the third finger as tightly as possible. Assessments will be conducted bilaterally, starting with the healthy side. The measurements will be repeated three times for each side, and the averages will be recorded in kg/f.

SECONDARY OUTCOMES:
Gross Grip Strength | 7 days
  For gross grip strength measurement, a hydraulic hand dynamometer (Baseline®, USA) will be used. The measurement will be conducted in the standard position specified by the American Society of Hand Therapists. In this position, the individual will sit on a chair with back support, with the elbow at 90 degrees of flexion and the wrist in a neutral position. The person will be asked to squeeze the dynamometer with maximum force. The measurement will be repeated three times, and the average will be recorded in kg/f.
Minnesota Manual Dexterity Test | 7 days
  The Minnesota Manual Dexterity Test (MMBT) consists of a board with 60 slots and 60 discs that fit into these slots. The test includes two subtests: the placing test and the turning test (Tesio, 2016).
  In the placing test, the discs are arranged at equal distances in front of the participant. The participant is then asked to pick up the disc closest to the board with their dominant hand and place it in the slot nearest to them. This continues by filling the columns and moving toward the non-dominant side. The time taken is recorded in seconds, from the moment the first disc is touched to when the last disc is placed in a slot. If a disc is dropped, the test continues without stopping the time, and the disc is picked up and placed again.
  The turning test begins with the discs already placed in the slots on the board. The participant turns the disc closest to the dominant hand on the top row with their non-dominant hand, progressing across the row toward the non-dominant side. They th
Moberg Pickup Test | 7 days
  The Moberg Pickup Test (MPT), developed by Moberg in 1958, is designed to evaluate the hand's ability to recognize small objects with and without visual input, as well as its functional sensory capacity. MPT assesses stereognosis and reflects motor performance (NG, 1999). In the test, the participant is asked to place 10 different objects (e.g., coins, nuts, a key, a screw, a nail, a paper clip, a safety pin, etc.) from the table into a box as quickly as possible. Measurements are taken four times: with and without visual input for both the dominant and non-dominant hand. The time is recorded in seconds, from the moment the participant touches the first object until the last object is placed in the box.
Purdue Pegboard Test | 7 days
  The Purdue Pegboard Test (PPT) assesses fine motor skills of the hand. The test begins by placing 25 pins, 20 washers, 40 collars, and 25 pins into four sections of the test board.
  For the dominant hand assessment, the participant is instructed, upon the command "start" from the administrator, to place the pins into the holes on the dominant side of the test board in sequence, without skipping any holes, within 30 seconds. The test time starts with the command, and the number of pins placed by the end is recorded on the assessment form.
  For the non-dominant hand assessment, the participant is instructed to place the pins on the board with the non-dominant hand, following the same procedure as with the dominant hand.
  For the bilateral assessment, the participant uses both hands simultaneously to place pins, beginning at the top hole. The test begins with the "start" command and ends after 30 seconds, with the number of pins placed recorded on the assessment form.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit Üniversitesi, Zonguldak, Turkey (Türkiye)